CLINICAL TRIAL: NCT04609345
Title: Prevalence of Ocular Surface Disease in Malaysian Glaucoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Santen Pharma Malaysia Sdn Bhd (Industry)
Responsible Party: Principal Investigator, Dr. Gan Eng Hui, Principal Investigator, International Specialist Eye Centre
Other Study IDs: CT20-004
Record Dates: First submitted 2020-10-20; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Primary Open-angle Glaucoma; Primary Angle-Closure Glaucoma; Pseudoexfoliation Glaucoma; Pigment Dispersion Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure; Exfoliation Syndrome; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, multi-centre, cross sectional observational study to determine the prevalence of ocular surface disease (OSD) in glaucoma patients, nationwide. The study also analyses sub group of OSD prevalence, stratified according to the treatment types (i.e. preserved, preservative-free, and combination of preservative-free and preserved eyedrops), and illustrates the patient perspective on OSD.

DETAILED DESCRIPTION:
For this prospective, multi-centre, cross sectional observational study, patients who attend routine eye examination at the medical institutions and who have been diagnosed with primary open-angle glaucoma, primary angle-closure glaucoma, pseudoexfoliation glaucoma, pigment dispersion glaucoma or ocular hypertension will be studied. The medical institutions are selected across different regions of Malaysia to assess the nationwide prevalence of OSD in glaucoma patients. The routine assessments include Corneal Evaluation, Tear Break-Up Time (TBUT), Hyperemia and Schirmer's test whereby the data from these assessments will be collected and analyzed. The study will also includes Symptom Evaluation and Questionnaire feedback.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age of 21 years or older and those who can provide informed consent.
* 2) On anti-glaucoma medications for >6 months
* 3) IOP ≤ 21 mm Hg in the study eye at the screening examination (under treatment)
* 4) If only one eye is eligible, it is to be evaluated. If both eyes are eligible, then the eye with a higher NEI score will be selected for evaluation.
* 5) A best-corrected visual acuity score of 6/36 on the Snellen Chart, or better in each eye.

Exclusion Criteria:

* 1) Those with secondary ocular hypertension or glaucoma
* 2) Those with severe visual field disorder (mean deviation of 20 dB or worse)
* 3) Those with a history of ocular surgeries (intraocular surgery including ocular laser treatment which may affect the patient's ocular surface condition) within 6 months prior to the study initiation.
* 4) Those with a history of glaucoma surgery
* 5) Those with a history of corneal refractive surgery
* 6) Those with severe dry eye associated with systemic disorders, or in need of drugs to treat dry eye
* 7) Those with ocular allergy, ocular infection or ocular inflammation
* 8) Those using eye drops for other ocular comorbidities
* 9) Those who need to use systemic or ophthalmic steroids (excluding topical skin steroidal ointment)
* 10) Female patients who are pregnant, nursing or lactating
* 11) Those who use contact lenses
* 12) Any corneal abnormality or other corneal comorbidity condition preventing reliable applanation tonometry
* 13) Those on oral antihistamine, antipsychotic or anti-depressant drugs.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attend routine eye examination at the medical institutions will be studied. The medical institutions are selected across different regions of Malaysia to assess the nationwide prevalence of OSD in glaucoma patients.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Fluorescein staining score (NEI/I) | 1 day
  The fluorescein stained area of the cornea and conjunctiva will be measured according to the National Eye Institute/Industry (NEI/I) method.
Tear Break-Up Time (TBUT) | 1 day
  The time (in seconds) until the tear film breaks and the corneal surface is exposed will be measured using a slitlamp microscope.
Hyperemia score | 1 day
  Bulbar and palpebral conjunctiva will be examined using the reference photographs and a 4-step scale. This 4-step scale is cited from the clinical evaluation criteria of Japanese Guideline for Allergic Conjunctival Diseases.
Schirmer's score | 1 day
  The test allows the water in tears to travel along the length of a paper test strip.

SECONDARY OUTCOMES:
Symptom Evaluation | 1 day
  Subjects will be evaluated for the presence of symptoms such as irritation/burning/stinging, foreign body sensation, tearing, itching and dry eye sensation.
Questionnaire feedback | 1 day
  Ocular Surface Disease Index (OSDI) patient questionnaire, Glaucoma QOL-15 questionnaire and Patient Experience Questionnaire (PEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Eng Hui Gan, Specialist, Principal Investigator — International Specialist Eye Centre (ISEC)

IPD SHARING:
Plan to Share IPD: Undecided
To be confirmed

REFERENCES:
- [Background] Harasymowycz P, Birt C, Gooi P, Heckler L, Hutnik C, Jinapriya D, Shuba L, Yan D, Day R. Medical Management of Glaucoma in the 21st Century from a Canadian Perspective. J Ophthalmol. 2016;2016:6509809. doi: 10.1155/2016/6509809. Epub 2016 Nov 8. PMID 27895937
- [Background] Jonas JB, Aung T, Bourne RR, Bron AM, Ritch R, Panda-Jonas S. Glaucoma. Lancet. 2017 Nov 11;390(10108):2183-2193. doi: 10.1016/S0140-6736(17)31469-1. Epub 2017 May 31. PMID 28577860
- [Background] Perez-Bartolome F, Martinez-de-la-Casa JM, Arriola-Villalobos P, Fernandez-Perez C, Polo V, Garcia-Feijoo J. Ocular Surface Disease in Patients under Topical Treatment for Glaucoma. Eur J Ophthalmol. 2017 Nov 8;27(6):694-704. doi: 10.5301/ejo.5000977. PMID 28497458
- [Background] Mathews PM, Ramulu PY, Friedman DS, Utine CA, Akpek EK. Evaluation of ocular surface disease in patients with glaucoma. Ophthalmology. 2013 Nov;120(11):2241-8. doi: 10.1016/j.ophtha.2013.03.045. Epub 2013 May 25. PMID 23714318
- [Background] Saade CE, Lari HB, Berezina TL, Fechtner RD, Khouri AS. Topical glaucoma therapy and ocular surface disease: a prospective, controlled cohort study. Can J Ophthalmol. 2015 Apr;50(2):132-6. doi: 10.1016/j.jcjo.2014.11.006. PMID 25863853
- [Background] Inoue K. Managing adverse effects of glaucoma medications. Clin Ophthalmol. 2014 May 12;8:903-13. doi: 10.2147/OPTH.S44708. eCollection 2014. PMID 24872675
- [Background] Ramli N, Supramaniam G, Samsudin A, Juana A, Zahari M, Choo MM. Ocular Surface Disease in Glaucoma: Effect of Polypharmacy and Preservatives. Optom Vis Sci. 2015 Sep;92(9):e222-6. doi: 10.1097/OPX.0000000000000542. PMID 25730335
- [Background] Garcia-Feijoo J, Sampaolesi JR. A multicenter evaluation of ocular surface disease prevalence in patients with glaucoma. Clin Ophthalmol. 2012;6:441-6. doi: 10.2147/OPTH.S29158. Epub 2012 Mar 22. PMID 22536034
- [Background] Ogawa Y, Kim SK, Dana R, Clayton J, Jain S, Rosenblatt MI, Perez VL, Shikari H, Riemens A, Tsubota K. International Chronic Ocular Graft-vs-Host-Disease (GVHD) Consensus Group: proposed diagnostic criteria for chronic GVHD (Part I). Sci Rep. 2013 Dec 5;3:3419. doi: 10.1038/srep03419. PMID 24305504
- [Background] Sencanic I, Gazibara T, Dotlic J, Stamenkovic M, Jaksic V, Bozic M, Grgurevic A. Validation of the Glaucoma Quality of Life-15 Questionnaire in Serbian language. Int J Ophthalmol. 2018 Oct 18;11(10):1674-1684. doi: 10.18240/ijo.2018.10.16. eCollection 2018. PMID 30364180
- [Background] Takamura E, Uchio E, Ebihara N, Ohno S, Ohashi Y, Okamoto S, Kumagai N, Satake Y, Shoji J, Nakagawa Y, Namba K, Fukagawa K, Fukushima A, Fujishima H; Japanese Society of Allergology. Japanese guideline for allergic conjunctival diseases. Allergol Int. 2011 Mar;60(2):191-203. doi: 10.2332/allergolint.11-RAI-0335. PMID 21636966
- [Background] Masumoto H, Tabuchi H, Yoneda T, Nakakura S, Ohsugi H, Sumi T, Fukushima A. Severity Classification of Conjunctival Hyperaemia by Deep Neural Network Ensembles. J Ophthalmol. 2019 Jun 2;2019:7820971. doi: 10.1155/2019/7820971. eCollection 2019. PMID 31275636
- [Background] Chan EW, Li X, Tham YC, Liao J, Wong TY, Aung T, Cheng CY. Glaucoma in Asia: regional prevalence variations and future projections. Br J Ophthalmol. 2016 Jan;100(1):78-85. doi: 10.1136/bjophthalmol-2014-306102. Epub 2015 Jun 25. PMID 26112871
- [Background] Holly FJ, Lamberts DW, Esquivel ED. Kinetics of capillary tear flow in the Schirmer strip. Curr Eye Res. 1982;2(1):57-70. doi: 10.3109/02713688208998380. PMID 7128183
- [Background] Miyake H, Kawano Y, Tanaka H, Iwata A, Imanaka T, Nakamura M. Tear volume estimation using a modified Schirmer test: a randomized, multicenter, double-blind trial comparing 3% diquafosol ophthalmic solution and artificial tears in dry eye patients. Clin Ophthalmol. 2016 May 13;10:879-86. doi: 10.2147/OPTH.S105275. eCollection 2016. PMID 27257372
- [Background] Bourne RRA, Kaarniranta K, Lorenz K, Traverso CE, Vuorinen J, Ropo A. Changes in ocular signs and symptoms in patients switching from bimatoprost-timolol to tafluprost-timolol eye drops: an open-label phase IV study. BMJ Open. 2019 Apr 2;9(4):e024129. doi: 10.1136/bmjopen-2018-024129. PMID 30944129
- See also: American Academy of Ophthalmology — https://www.aao.org/image/neiindustry-grading-system